CLINICAL TRIAL: NCT05200988
Title: A Phase 2 Clinical Study to Assess Efficacy of Induction Ipilimumab/Nivolumab to Spare the Bladder in Urothelial Bladder Cancer
Brief Title: Checkpoint Inhibition and Chemoradiotherapy as Bladder Sparing Treatment in UC
Acronym: Indi-Blade
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21IDB
Record Dates: First submitted 2021-10-14; First posted 2022-01-21 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, phase 2 clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction with heckpoint inhibition followed by consolidative chemoradiation (Experimental): Checkpoint inhibition and chemoradiation
  Interventions: Drug: Ipilimumab + nivolumab

INTERVENTIONS:
Drug: Ipilimumab + nivolumab — Induction with immune checkpoint blockade: ipilimumab 3mg/kg on day 1, pilimumab 3mg/kg plus nivolumab 1mg/kg on day 22, and nivolumab 3mg/kg on day 43
  Response evaluation after the last cycle of checkpoint inhibition.
  Chemoradiation will start 10-12 weeks after start of checkpoint inhibition according to the following scheme:
  * Mitoycine C (12mg/m2) on the first day of radiotherapy, followed by either 5-fluorouracil intravenously (500mg/m2) five days a week during week one and four of radiation, or oral capecitabin (2x825mg/m2) every day during the radiation period
  * Radiation with a preference for a four-week schedule, in which 55 Gy will be administered using intensity modulated radiation therapy
  Other Names: Yervoy; Opdivo

SUMMARY:
This is a single-armed, multicenter, non-blinded phase 2 study to assess efficacy of induction ipilimumab + nivolumab followed by chemoradiation to spare the bladder in urothelial bladder cancer.

DETAILED DESCRIPTION:
This is a phase 2 study in which fifty adult patients with cT2-4aN0-2 urothelial bladder cancer, who are amenable for chemoradiation, will be included. Lymph nodes should be amenable for inclusion into the radiation field.

Included patients will be treated with three cycles of checkpoint inhibition: ipilimumab 3mg/kg on day 1, ipilimumab 3 mg/kg plus nivolumab 1 mg/kg on day 22, and nivolumab 3 mg/kg on day 43.

Response of this induction therapy will be evaluated by cystoscopy, mpMRI and a CT scan.

Patients will then be treated by radiation to the bladder and involved nodes, in combination with mitomycine C (day 1, 12 mg/m2, maximum dose of 20 mg) and either daily capecitabin or intravenous 5-FU in week 1 and 4. Radiotherapy will be delivered using Volumetric Modulated Arc Therapy delivering a dose of 50Gy to the whole bladder with a simultaneous tumor boost of 60Gy to the tumor bed.

The primary endpoint is efficacy, defined as bladder-intact event-free survival (BI-EFS). Events consist of death by any cause; muscle-invasive, upper urinary tract, nodal or distant recurrence, cystectomy, or switch to cisplatin-based chemotherapy.

The first evaluation after completion of chemoradiation will be after three months. Further follow-up visits will take place 6, 12, 18, 24, 30, and 36 months after completion of chemoradiation. During these visits, focused physical examination, cystoscopy and a CT chest-abdomen will be performed, combined with registration of treatment-related adverse events and a questionnaire for evaluating QoL, bladder function and long-term effects of immunotherapy on QoL.

Key secondary endpoints are overall survival (OS), recurrence-free survival (RFS), feasibility to proceed to chemoradiation, safety, QoL, and bladder function.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Age ≥ 18 years
3. Patients with cT2-4aN0-2M0 urothelial bladder cancer, who are amendable for chemoradiation and who are seeking an alternative to radical cystectomy and/or patients who are medically unfit for surgery.
4. Lymph nodes should be amenable for inclusion into the radiation field.
5. World Health Organization (WHO) performance Status 0 or 1.
6. Urothelial cancer is the dominant histology (>70%). A small cell component is not allowed.
7. Formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks from diagnostic TUR available.
8. Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥1.0x109/L, Platelets ≥100 x109/L, Hemoglobin ≥5.5 mmol/L, GFR>30 ml/min as per Cockcroft-Gault formula, AST ≤ 2.5 x ULN, ALT ≤2.5 x ULN, Bilirubin ≤1.5 X ULN
9. Negative pregnancy test (βHCG in urine or blood) for female patients of childbearing potential within 2 weeks prior to day 1 of start immunotherapy.
10. Highly effective contraception for both male and female subjects if the risk of conception exists. Female patients of childbearing potential must comply with contraception methods as requested by the study protocol.

Exclusion Criteria:

1. Previous pelvic irradiation
2. Upper tract urothelial cancer
3. Extensive carcinoma in situ (CIS) of the bladder
4. Bilateral hydronephrosis
5. Previous intravenous chemotherapy for bladder cancer
6. Contra-indication to one of the study treatment components, or mpMRI
7. Subjects with active autoimmune disease in the past 2 years. Patients with diabetes mellitus, properly controlled hypothyroidism or hyperthyroidism, vitiligo, psoriasis or other mild skin disease can still be included.
8. Documented history of severe autoimmune disease (e.g. inflammatory bowel disease, myasthenia gravis).
9. Prior CTLA-4 or PD-(L)1 -targeting immunotherapy.
10. Known history of Human Immunodeficiency Virus, active tuberculosis, or other active infection requiring therapy at the time of inclusion.
11. Positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA)
12. Underlying medical conditions that, in the investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of adverse events
13. Medical condition requiring the use of immunosuppressive medications, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) will be allowed.
14. Use of other investigational drugs four weeks before study drug administration
15. Malignancy, other than urothelial cancer, in the previous 2 years, with a high chance of recurrence (estimated >10%). Patients with low risk prostate cancer (defined as Stage T1/T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL) who are treatment-naive and undergoing active surveillance are eligible.
16. Pregnant and lactating female patients.
17. Major pelvic surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
18. Severe infections within 2 weeks prior to enrolment in the study including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2027-09-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy defined as bladder-intact event-free survival (BI-EFS) | From initiation of study drug until event, defined as described above, whichever comes first. Patients without an event are censored at time of last cystoscopy/last CT scan. Assessed at primary analysis and subsequently at a minimum of 3yrs follow-up.
  Events are defined as death by any cause, muscle-invasive, upper urinary tract, nodal or distant recurrence, cystectomy, or switch to cisplatin-based chemotherapy.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | From start of therapy until one of the events mentioned above, whichever comes first. RFS will be assessed at the primary analysis and subsequently at a minimum of 3 years follow-up for all patients
  RFS is defined as time from start of therapy until the following events: muscle-invasive bladder or upper urinary tract recurrence, locoregional or distant metastases, switch to cisplatin-based chemotherapy or death by any cause.
Overall survival (OS) | From date of enrollment until date of death. OS will be assessed at the primary analysis and subsequently at a minimum of 3 years follow-up for all patients.
  OS is defined as the time between the date of enrollment and the date of death.
Feasibility to proceed to chemoradiation (CRT) | From the initiation of the study drug untill the the start of CRT
  Percentage of patients able to proceed to CRT
Change in patient reported outcome regarding quality of life (QoL) | From screening until two years after finalizing chemoradiation
  QoL will be assessed using the EORTC QLQ-C30 and an unvalidated immunotherapy-related QoL questionnaire developed by and used in the Netherlands Cancer Institute. These will be provided to evaluate changes from baseline in QoL and evaluate long-term effects of immunotherapy on QoL using both multi-item scale and single-item scales. A graph showing the change from baseline to three timepoints will be reported: 56 ±7 days after treatment initiation and at 3, 6, 12,18 and 24 months after finalizing chemoradiotherapy.
Patient reported outcome regarding bladder function | From screening until two years after finalizing chemoradiation
  Questionnaires for bladder function (EORTC-QLQ-BLM30)will be provided, resulting in a score on a four point scale. A graph showing the change from baseline to six timepoints will be reported: 56 ±7 days after treatment initiation and at 3, 6, 12,18 and 24 months after finalizing chemoradiotherapy.

OTHER OUTCOMES:
Radiological tumor evaluation by mpMRI | mpMRI assessments will be done at baseline and at 56 ±7 days after treatment initiation. BI-EFS, RFS and OS will be determined as mentioned above and collected at the moment of primary analysis.
  Tumor evaluation by AI based radiological assessment of pre- and on-treatment mpMRI will be established to identify nonresponding patients. BI-EFS, RFS and OS will be compared for the binary outcome mpMRI response vs nonresponse.
Translational | TMB and PD-L1 will be determined on baseline tissue. BI-EFS, RFS and OS will be determined as mentioned above.
  BI-EFS, RFS and OS will be compared between patients with Tumor mutational burden (TMB) >median vs <median.
  BI-EFS, RFS and OS will be compared between patients with PD-L1 high tumors versus patients with PD-L1 low tumors.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Antoni van Leeuwenhoek ziekenhuis, Amsterdam
  - Erasmus Medical Center, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht

REFERENCES:
- [Derived] Stockem CF, Mellema JJJ, van Rhijn BWG, Boellaard TN, van Montfoort ML, Balduzzi S, Boormans JL, Franckena M, Meijer RP, Robbrecht DGJ, Suelmann BBM, Schaake EE, van der Heijden MS. Induction therapy with ipilimumab and nivolumab followed by consolidative chemoradiation as organ-sparing treatment in urothelial bladder cancer: study protocol of the INDIBLADE trial. Front Oncol. 2023 Aug 29;13:1246603. doi: 10.3389/fonc.2023.1246603. eCollection 2023. PMID 37711193